CLINICAL TRIAL: NCT03024047
Title: Cohort Description of Younger With AV-block
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: DAN-BLOCK_Study1
Record Dates: First submitted 2017-01-04; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Atrioventricular Block; Progressive Cardiac Conduction Defect; Genetic Disease
MeSH Terms: conditions — Atrioventricular Block; Bundle-Branch Block; Genetic Diseases, Inborn

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Pacemaker

SUMMARY:
Background:

Disturbances of the heart's atrioventricular conduction - AV-block - may show by shortness of breath, fainting or sudden death. If AV-block is diagnosed in time pacemaker therapy may be lifesaving.

AV-block in younger can be seen along with structural or ischemic heart disease, congenital heart disease (incl. congenital AV-block) storage disorders, specific muscle diseases, sarcoidosis, Borrelia infection or drug intoxication. AV-block in younger can also be seen in conditions, primarily localized to the AV-node without other cardiac disease at diagnosis.

This form of AV-block is often hereditary and can be seen in families where relatives have another types of heart disease in form of fore example, cardiomyopathy, ion channel disease or sudden death. The different forms of presentation are due to the same gene mutation being expressed differently within the same family. Thus, early onset of AV-block (<50 years) may indicate hereditary AV-conduction disorder but it can also be the first manifestation of severe ion channel disease or cardiomyopathy.

Denmark has annually over 50 individuals <50 years treated with pacemaker due to advanced AV-block. There have been no overall figures regarding the causes of advanced AV-block, and therefore no systematic approach to diagnosing this group of patients. Furthermore, the prevalence of individuals with a genetic cause of AV-block is unknown and presumably an often overlooked diagnosis among younger patients with advanced AV-blok. There are no data on disease progression after diagnosis, and therefore there is no evidence-based knowledge about how these patients should be followed after diagnosis.

With modern gene technology, a range of new, yet unknown genes with potentially pathogenic mutations is likely to be identified. Identification of such genes, and the development of a strategy for systematic approach to diagnose younger patients with AV-block, will enable presymptomatic genetic screening of relatives and implementation of evidence-based, preventive treatment with pacemaker and/or medical treatment for heart failure based on a specific genetic predisposition for development of AV-block with or without heart failure.

Hypotheses:

In a significant proportion of younger patients with advanced AV-block the underlying cause is unknown.

Objective:

To investigate the prevalence and causes of advanced AV-block in younger patients in Denmark and describe the current diagnostics.

Method:

The study is a cross sectional study. The patients for this study are identified from Danish Pacemaker and ICD Register. The investigators will review medical records and obtain clinical information and test results (see detailed description).

Perspectives:

This study is the first part of a large study of AV-block in younger patients in Denmark. The overall goal, is to increase knowledge about the causes of and disease progression after the diagnosis of advanced AV-block in young patients which could lead to a significant improvement in the treatment of this patient group and may lead to a customized choice of pacemaker type in the future and perhaps additional medical treatment in this patient group. This could potentially lead to a reduction in both their morbidity mortality.

DETAILED DESCRIPTION:
Method:

The following covariates will be reported.

Date of diagnosis of AV-block:

The date of diagnosis is defined as the day the physician diagnoses the AV-block. E.g. if the patient has a Holter monitoring performed, the date of diagnosis is the dag the monitoring is reviewed.

Reported as: Day-month-year

Comorbidity at day of first pacemaker implant:

Registered as one or more of the following:

1. Diabetes
2. Hypertension
3. Hypercholesterolemia
4. Heart failure
5. Atrial fibrillation or flutter
6. Ischemic heart disease
7. Sarcoidosis
8. Connecting tissue disorder
9. Other

Smoking status at day of first pacemaker implant:

Registered as: Current, former, never

Device selected at first pacemaker implant:

Registered as: DDD, CTR, etcetera

Genetic investigation:

Is there performed genetic investigation due to the finding of AV-block? Investigation must be initiated maximum 4 weeks after day of first pacemaker implant.

Registered as: y/n.

Date of first pacemaker implant:

Registered as: Day-month-year

Implant sight

ECG 12 description:

ECG 12 must be taken maximum one week before day of first pacemaker implant Registered as: Bpm., RBBB y/n, LBBB y/n, PR in msec, QRS in msec, QT in msec, QTc in msec (Frederica)

Implant indication:

Registered as one of following:

1. First-degree atrioventricular block with symptoms
2. Mobitz type 1 with symptoms
3. Mobitz type 2
4. Advanced second-degree atrioventricular block
5. Third-degree atrioventricular block
6. Unknown The most malignant is chosen and it is reported if it is intermittent or persistent.

Symptoms:

Registered as one or more of following:

1. Dyspnoea
2. Fatigue
3. Malaise
4. Dizziness
5. Syncope
6. Angina
7. Cardiac arrest
8. No symptoms

Echocardiography:

Performed maximum two weeks before day of first pacemaker implant The reported values are what the echocardiographer describes.

Registered as:

LVEF in % (values over 60% is reported as >60 %) Hypertrophy of LV y/n Dilatation of LV y/n Dilatation of LA y/n Valvular disease/artificial valve y/n

Coronary angiography:

At day of first pacemaker implant +/- 4 weeks

Registered as:

Normal y/n Significantly disease on LAD y/n Significantly disease on RCA y/n Significantly disease on CX y/n Significantly disease = leading to CABG, PCI or antithrombotic treatment

ELIGIBILITY:
Inclusion Criteria:

* All patients in Denmark
* Treated with pacemaker due to AV-block
* Implanted for the first time between 01.01.1996 - 31.12.2015
* Age at implantation <50 years

Exclusion Criteria:

* Non

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients in Denmark with AV-block who were treated with pacemaker for the first time between 01.01.1996 - 31.12.2015 with age at implantation <50 years will be included in the study (n=1,255 patients).
Sampling Method: Probability Sample
Enrollment: 1255 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of structural heart disease as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of ischemic heart disease as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of congenital heart disease as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of congenital AV-block | 01.01.1996 - 31.12.2015
Prevalence of muscular dystrophy as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of sarcoidosis as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of lyme disease as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of genetic cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of complications to operation as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of complications to radio frequency ablation as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of endocarditis as cause of AV-block | 01.01.1996 - 31.12.2015
Prevalence of unknown cause of AV-block | 01.01.1996 - 31.12.2015

CONTACTS AND LOCATIONS:
Locations (1):
- Department of cardiology, Research, Aarhus University Hospital, Denmark, Aarhus, Denmark